CLINICAL TRIAL: NCT07214935
Title: A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of Evobrutinib on the QTc (Corrected QT) Interval in Healthy Adult Participants
Brief Title: A TQT Study of Effect of M2951 on Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MS200527_0070; 2022-002664-78 (EudraCT Number)
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Healthy
Keywords: M2951; Bruton's Tyrosine Kinase; Cardiac Repolarization
MeSH Terms: interventions — Moxifloxacin; evobrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants will receive one of the four interventions in a sequence decided at randomization.
  Interventions: Drug: Placebo matched to M2951; Drug: Moxifloxacin; Drug: M2951 Low Dose; Drug: M2951 High Dose
- Treatment Sequence 2 (Experimental): Participants will receive one of the four interventions in a sequence decided at randomization.
  Interventions: Drug: Placebo matched to M2951; Drug: Moxifloxacin; Drug: M2951 Low Dose; Drug: M2951 High Dose
- Treatment Sequence 3 (Experimental): Participants will receive one of the four interventions in a sequence decided at randomization.
  Interventions: Drug: Placebo matched to M2951; Drug: Moxifloxacin; Drug: M2951 Low Dose; Drug: M2951 High Dose
- Treatment Sequence 4 (Experimental): Participants will receive one of the four interventions in a sequence decided at randomization.
  Interventions: Drug: Placebo matched to M2951; Drug: Moxifloxacin; Drug: M2951 Low Dose; Drug: M2951 High Dose

INTERVENTIONS:
Drug: Placebo matched to M2951 — Participants will receive single oral dose of placebo matched to M2951 in either of study periods (period 1 or period 2 or period 3 or period 4) under fasted conditions.
Drug: Moxifloxacin — Participants will receive single oral dose of moxifloxacin in either of study periods (period 1 or period 2 or period 3 or period 4) under fasted conditions.
Drug: M2951 Low Dose — Participants will receive single oral low dose of M2951 in either of study periods (period 1 or period 2 or period 3 or period 4) under fasted conditions.
  Other Names: Evobrutinib; MSC2364447C
Drug: M2951 High Dose — Participants will receive single oral high dose of M2951 in either of study periods (period 1 or period 2 or period 3 or period 4) under fasted conditions.
  Other Names: Evobrutinib; MSC2364447C

SUMMARY:
The purpose of this study is to assess potential effects of M2951 on cardiac repolarization (i.e. prolongation of QT interval).

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as determined by medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection, or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Participants have a body weight within 50.0 and 100.0 kilograms (kg) (inclusive) and body mass index (BMI) within the range 19.0 and 30.0 kilograms per square meter (kg/m^2) (inclusive)
* Participants are stable nonsmokers for at least 3 months preceding the first administration of study intervention

Exclusion Criteria:

* Participants with history or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue, psychiatric (due to rare risk of hallucinations, agitation, and activation of psychosis), and other diseases or disorders, and epilepsy, as determined by medical evaluation
* Participants with diagnosis of hemochromatosis, Wilson´s disease, alpha 1 antitrypsin deficiency, or any other chronic liver disease including Gilbert's disease will be excluded from the study. Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to the first administration of study intervention
* Participants with history of any malignancy
* Participants with history of seizures
* Participants with history of pharmacologically treated psychiatric disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Participants received single oral dose of Placebo on Day 1 in fasted state in Period 1, followed by single oral dose of moxifloxacin 400 mg tablet on Day 8 in fasted state in Period 2, followed by 45 mg single dose of oral solution of evobrutinib in fasted state on Day 15 in Period 3, and 225mg single dose of oral solution of evobrutinib in fasted state on Day 22 in period 4. A washout period of 7 days was maintained between 4 treatment periods
- Sequence 2: Participants received single oral dose of moxifloxacin 400 mg tablet on Day 1 in fasted state in Period 1, followed by single oral dose of Evobrutinib 225 mg solution on Day 8 in fasted state in Period 2, followed by single oral dose of Placebo in fasted state on Day 15 in Period 3, and 45 mg of dose of single oral solution of evobrutinib in fasted state on Day 22 in period 4. A washout period of 7 days was maintained between 4 treatment periods
- Sequence 3: Participants received single oral dose of evobrutinib 45 mg solution on Day 1 in fasted state in Period 1, followed by single oral dose of Placebo on Day 8 in fasted state in Period 2, followed by single oral dose of 225 mg evobrutinib solution in fasted state on Day 15 in Period 3, and 400 mg of dose of single oral tablet of moxifloxacin in fasted state on Day 22 in period 4. A washout period of 7 days was maintained between 4 treatment periods
- Sequence 4: Participants received single oral dose of evobrutinib 225 mg solution on Day 1 in fasted state in Period 1, followed by single oral dose of 45 mg evobrutinib solution on Day 8 in fasted state in Period 2, followed by single oral dose of 400 mg moxifloxacin tablet in fasted state on Day 15 in Period 3, and single oral dose of Placebo in fasted state on Day 22 in period 4. A washout period of 7 days was maintained between 4 treatment periods
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 9 | 9 | 9
Completed | 7 | 7 | 8 | 8
Not Completed | 2 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Participant did not meet all eligibility criteria, ADMISSION DRUG SCREEN POSITIVE | 1 | 0 | 0 | 0
Not completed — Participant discontinued prior to first dosing | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (7.5) | 36 (10.4) | 41 (8.6) | 40 (11.3) | 41 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 8
  Male | 6 | 7 | 7 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 9 | 8 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 8 | 8 | 8 | 8 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Placebo-corrected Change From Baseline in Corrected QT Interval by Fridericia' Formula (QTcF) for Evobrutinib
Description: A linear mixed-effects model was used to analyze the relationship between evobrutinib and MSC2729909A concentrations and ΔQTc. Based on this model, drug-induced ΔΔQTc and its two-sided 90% CI was predicted over the clinical concentration range and at concentrations corresponding to the observed geometric mean Cmax following administration of 45 mg and 225 mg evobrutinib. The higher geometric mean Cmax calculated based on the PK and ECG Analysis Sets was considered.
Time Frame: Baseline and from 1 hour before any administration until 24 hours post-administration at the following timepoints: -1-hour, 5 min, 10 min, 20 min, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours
Population: The ECG analysis set includes all participants who had a baseline Holter ECG in triplicate and at least one post baseline Holter ECG in triplicate with a time-matched concentration
Measure: Geometric Mean (95% Confidence Interval); unit: milliseconds
Groups:
- Evobrutinib 45mg: Participants received single oral dose of Evobrutinib 45 milligram (mg) in treatment period 1, 2, 3 or 4 under fasted condition
- Evobrutinib 225mg: Participants received single oral dose of Evobrutinib 225 mg in treatment period 1, 2, 3 or 4 under fasted condition
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg
Number analyzed (Participants) | 31 | 32
milliseconds | -1.62 [-2.15 to -1.09] | -2.28 [-3.63 to -0.93]

2. Secondary Outcome: Placebo-corrected Change From Baseline in Corrected QT Interval by Fridericia' Formula (QTcF) for Moxifloxacin
Description: A linear mixed-effects model was used to analyze the relationship between moxifloxacin concentrations and ΔQTc. Based on this model, drug-induced ΔΔQTc and its two-sided 90% CI was predicted. The higher geometric mean Cmax calculated based on the PK and ECG Analysis Sets was considered.
Time Frame: From 1 hour before any administration until 24 hours post-administration at the following timepoints: -1-hour, 5 min, 10 min, 20 min, 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hours
Population: All participants who had a baseline Holter ECG in triplicate and at least one post baseline Holter ECG in triplicate with a time-matched concentration.
Measure: Geometric Mean (95% Confidence Interval); unit: milliseconds
Groups:
- Moxifloxacin 400mg: Participants received single oral dose of Moxifloxacin 400 mg treatment period 1, 2, 3 or 4 under fasted condition
Arm/Group | Moxifloxacin 400mg
Number analyzed (Participants) | 32
milliseconds | 12.2 [10.3 to 14.1]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment.Therefore, an AE can be any unfavorable and unintended sign (including an abnormallaboratory finding), symptom, or disease temporally associated with the use of amedicinal product, regardless if it is considered related to the medicinal product.Serious AE: AE that resulted in any of the following outcomes: death; life threatening;persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization;congenital anomaly/birth defect. TEAEs are defined as AEs that were reported orworsened on or after start of study drug dosing through the Safety Follow-up Visit.TEAEs included both serious TEAEs and non-serious TEAEs. Treatment related AEs:reasonably related to the study drug/study treatment.
Time Frame: Up to 3 months
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Moxifloxacin 400mg: Participants received single oral dose of Moxifloxacin 400 mg in treatment period 1, 2, 3 or 4 under fasted condition
- Placebo: Participants received single oral solution of placebo in treatment period 1, 2, 3 or 4 under fasted condition
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
Participants | 8 | 5 | 5 | 8

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on Severity
Description: Severity of adverse events (AE) were assessed by the investigator. The Investigator assessed the intensity of each AE and SAE reported during the study and assigned it to 1 of the following categories:
  1. Mild: A type of adverse event that is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. 2. Moderate: A type of adverse event that is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. 3. Severe: A type of adverse event that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Number of participants with severe adverse events were reported.
Time Frame: Up to 3 months
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Evobrutinib 45mg: Participants received single oral dose of Evobrutinib 45 mg in treatment period 1, 2, 3 or 4 under fasted condition
- Evobrutinib 225mg: Participants received single oral dose of Evobrutinib 225 mg n treatment period 1, 2, 3 or 4 under fasted condition
- Moxifloxacin 400mg: Participants received single oral dose of Moxifloxacin 400 mg n treatment period 1, 2, 3 or 4 under fasted condition
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities From Baseline in Safety Laboratory Tests
Description: The laboratory measurements included hematology, blood chemistry and urinalysis. Number of participants with clinically significant abnormalities from baseline were reported. Clinically Significance was decided by investigator.
Time Frame: Up to Day 29
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Evobrutinib 45mg: Participants received single oral dose of Evobrutinib 45 mg in Period 1, 2, 3 or 4 under fasted condition
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities From Baseline in Vital Signs
Description: Vital sign assessment included blood pressure, pulse rate, body temperature and respiration (frequency per minute). Number of participants with clinically significant abnormalities in vital signs were reported. Clinically significance was decided by investigator.
Time Frame: Up to Day 29
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Electroencephalogram (EEG) and Electrocardiogram (ECG) Findings
Description: The 12-lead ECG recordings were obtained after 5 minutes of rest in a semi-supine position. ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, QT and QTc intervals. Number of participants with clinically significant abnormalities were reported. Clinically significance was decided by investigator.
Time Frame: Up to Day 29
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Blood-Concentration Time Curve From Time Zero to 24 Hours Post-Dose (AUC 0-24) of Evobrutinib
Description: AUC from time zero to 24 hours post dose, calculated using the mixed log linear trapezoidal rule (linear up, log down) using the nominal dosing interval.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: The PK Analysis Set was a subset of the SAF, and the PK population included all participants: who had completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results and with adequate study intervention compliance and with evaluable PK data, i.e. no missing values for primary endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg
Number analyzed (Participants) | 30 | 30
hour*nanogram/milliliter | 249 (38.4) | 1420 (37.5)

9. Secondary Outcome: Area Under the Plasma-Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC 0-inf) of Evobrutinib
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at t last, as estimated using the linear regression from lambda (λ)z determination.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg
Number analyzed (Participants) | 30 | 30
h*ng/mL | 248 (38.4) | 1420 (37.5)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Evobrutinib
Description: Cmax is the maximum observed plasma concentration. Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg
Number analyzed (Participants) | 30 | 30
ng/mL | 123 (45.8) | 670 (51.3)

11. Secondary Outcome: Time to Reach Maximum Blood Concentration (Tmax) of Evobrutinib
Description: Time to reach the maximum blood concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg
Number analyzed (Participants) | 30 | 30
hours | 0.500 [0.267 to 2.02] | 0.500 [0.250 to 2.03]

12. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Evobrutinib
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg
Number analyzed (Participants) | 30 | 30
hours | 1.32 (22.7) | 2.09 (33.8)

13. Secondary Outcome: Area Under the Blood-Concentration Time Curve From Time Zero to 24 Hours Post-Dose (AUC 0-24) Of Moxifloxacin
Description: as for outcome 8
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Moxifloxacin 400mg
Number analyzed (Participants) | 30
h*ng/mL | 19600 (19.6)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Moxifloxacin
Description: Cmax is the maximum observed plasma concentration. Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Moxifloxacin 400mg
Number analyzed (Participants) | 30
ng/mL | 2000 (30.3)

15. Secondary Outcome: Area Under the Plasma-Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC 0-inf) of Moxifloxacin
Description: as for outcome 9
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Moxifloxacin 400mg
Number analyzed (Participants) | 30
h*ng/mL | 24900 (19.8)

16. Secondary Outcome: Time to Reach Maximum Blood Concentration (Tmax) of Moxifloxacin
Description: Time to reach the maximum blood concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose up to 24 hours post-dose on Days 1, 8, 15, and 22
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Moxifloxacin 400mg
Number analyzed (Participants) | 30
hours | 1.50 [0.250 to 4.00]

17. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: ECG Mean Heart Rate
Description: The effect of evobrutinib on baseline-corrected measurements of Heart rate was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: Baseline, and post-dose at 15 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 16 hours, and 24 hours
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
beats/min
  Baseline | 58.1 (8.38) | 58.6 (7.38) | 58.7 (7.90) | 57.9 (7.61)
  15 Minutes Post-dose | 0.6 (3.26) | 1.3 (3.83) | 0.0 (2.58) | 0.8 (2.65)
  30 Minutes Post-dose | 0.0 (3.43) | 0.2 (3.26) | 1.6 (3.57) | 0.7 (2.98)
  1 Hour Post-dose | 1.7 (3.68) | 1.0 (4.00) | 2.6 (3.80) | 3.2 (4.10)
  1.5 Hour Post-dose | 1.7 (3.26) | 1.1 (3.60) | 3.0 (3.48) | 3.9 (4.03)
  2 Hour Post-dose | 0.6 (3.10) | 1.4 (2.21) | 3.6 (4.76) | 2.8 (3.05)
  2.5 Hour Post-dose | 0.4 (4.04) | 0.7 (3.73) | 1.9 (4.22) | 1.2 (3.64)
  3 Hour Post-dose | -0.4 (4.43) | -0.0 (3.28) | 2.4 (3.63) | 1.9 (4.13)
  4 Hour Post-dose | 0.8 (3.67) | 0.8 (3.54) | 2.7 (6.52) | 2.7 (4.03)
  6 Hour Post-dose | 6.6 (6.42) | 6.1 (4.85) | 7.8 (4.84) | 9.3 (5.53)
  8 Hour Post-dose | 4.2 (5.85) | 2.3 (5.29) | 5.5 (4.24) | 5.2 (5.30)
  12 Hour Post-dose | 1.3 (5.36) | -0.1 (4.63) | 2.6 (5.62) | 0.7 (4.75)
  16 Hour Post-dose | 3.5 (5.91) | 2.1 (5.73) | 4.6 (5.25) | 5.6 (5.16)
  24 Hour Post-dose | 6.0 (7.88) | 2.6 (5.62) | 4.3 (5.38) | 5.3 (5.69)

18. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: RR Interval
Description: The effect of evobrutinib on baseline-corrected measurements of RR interval was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: as for outcome 17
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
milliseconds
  Baseline | 1057.4 (146.41) | 1044.0 (139.39) | 1043.4 (144.03) | 1056.1 (140.61)
  15 Minutes Post-dose | -14.8 (60.09) | -24.4 (63.48) | 0.6 (45.64) | -13.8 (54.73)
  30 Minutes Post-dose | -4.2 (65.10) | -4.9 (55.65) | -26.6 (66.04) | -11.3 (48.52)
  1 Hour Post-dose | -30.2 (72.81) | -17.0 (60.28) | -40.3 (62.87) | -47.3 (58.95)
  1.5 Hour Post-dose | -34.4 (65.46) | -17.2 (59.43) | -52.5 (59.00) | -66.0 (78.10)
  2 Hour Post-dose | -14.0 (57.06) | -26.2 (40.34) | -65.0 (81.34) | -49.9 (57.51)
  2.5 Hour Post-dose | -10.8 (69.18) | -10.6 (70.27) | -37.4 (79.84) | -18.8 (65.83)
  3 Hour Post-dose | 0.2 (80.54) | -1.8 (65.55) | -45.2 (74.46) | -31.8 (81.31)
  4 Hour Post-dose | -20.1 (67.37) | -15.9 (61.57) | -48.1 (99.08) | -44.6 (71.37)
  6 Hour Post-dose | -112.1 (115.18) | -101.1 (94.08) | -127.3 (89.62) | -146.5 (94.86)
  8 Hour Post-dose | -74.0 (95.45) | -38.8 (95.45) | -97.8 (83.82) | -83.7 (88.55)
  12 Hour Post-dose | -24.8 (94.78) | 1.4 (89.18) | -47.3 (103.93) | -15.7 (93.15)
  16 Hour Post-dose | -61.3 (98.99) | -39.9 (105.20) | -83.3 (99.08) | -94.7 (84.41)
  24 Hour Post-dose | -98.8 (127.77) | -42.6 (106.76) | -74.0 (101.40) | -85.1 (88.69)

19. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: QT Interval
Description: The effect of evobrutinib on baseline-corrected measurements of QT interval was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: as for outcome 17
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
milliseconds
  Baseline | 395.8 (28.44) | 393.2 (27.84) | 394.5 (26.29) | 396.4 (27.77)
  15 Minutes Post-dose | -0.1 (6.99) | -1.5 (6.70) | 0.1 (6.34) | 1.2 (8.39)
  30 Minutes Post-dose | 0.6 (8.71) | -0.5 (5.61) | -1.7 (7.29) | 0.1 (7.44)
  1 Hour Post-dose | -5.2 (8.86) | -2.8 (7.99) | 3.6 (10.74) | -5.0 (9.08)
  1.5 Hour Post-dose | -8.0 (8.12) | -6.0 (8.93) | 3.2 (10.41) | -8.2 (11.75)
  2 Hour Post-dose | -4.3 (7.63) | -6.9 (6.62) | 3.5 (13.02) | -7.4 (10.21)
  2.5 Hour Post-dose | -4.5 (9.55) | -5.4 (9.46) | 5.5 (11.71) | -4.1 (10.14)
  3 Hour Post-dose | -3.5 (10.58) | -3.6 (9.31) | 5.3 (12.19) | -6.0 (12.45)
  4 Hour Post-dose | -5.7 (9.95) | -4.4 (10.67) | 2.4 (16.10) | -7.8 (10.66)
  6 Hour Post-dose | -19.2 (15.98) | -16.9 (13.10) | -13.6 (13.12) | -22.3 (14.43)
  8 Hour Post-dose | -13.7 (13.06) | -11.3 (13.33) | -8.2 (12.25) | -14.2 (12.80)
  12 Hour Post-dose | -2.7 (14.12) | -0.7 (13.23) | 1.4 (14.28) | -1.7 (12.04)
  16 Hour Post-dose | -4.1 (14.04) | -0.8 (15.15) | -0.9 (13.19) | -8.5 (13.26)
  24 Hour Post-dose | -16.3 (18.95) | -9.5 (13.66) | -8.5 (13.92) | -15.8 (12.30)

20. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: QTcF Interval
Description: The effect of evobrutinib on baseline-corrected measurements of QTcF was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: as for outcome 17
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
milliseconds
  Baseline | 389.4 (18.08) | 388.4 (17.88) | 389.8 (17.28) | 390.0 (17.58)
  15 Minutes Post-dose | 1.6 (4.50) | 1.6 (4.66) | -0.1 (3.91) | 2.8 (3.75)
  30 Minutes Post-dose | 0.8 (5.08) | 0.0 (3.77) | 1.8 (5.90) | 1.6 (4.26)
  1 Hour Post-dose | -1.2 (4.49) | -0.7 (4.62) | 8.8 (7.14) | 1.3 (5.16)
  1.5 Hour Post-dose | -3.7 (4.50) | -3.8 (5.04) | 9.8 (8.09) | 0.2 (5.46)
  2 Hour Post-dose | -2.7 (3.77) | -3.6 (3.98) | 11.7 (7.92) | -1.1 (5.61)
  2.5 Hour Post-dose | -3.3 (5.26) | -3.9 (4.87) | 10.0 (6.33) | -1.7 (4.52)
  3 Hour Post-dose | -3.7 (5.89) | -3.4 (4.64) | 10.8 (5.78) | -1.9 (5.29)
  4 Hour Post-dose | -3.3 (5.34) | -2.4 (5.80) | 8.4 (7.03) | -2.0 (5.54)
  6 Hour Post-dose | -5.0 (7.51) | -4.0 (7.07) | 3.0 (8.24) | -3.4 (7.51)
  8 Hour Post-dose | -4.5 (5.64) | -6.2 (7.41) | 4.2 (8.00) | -3.4 (7.85)
  12 Hour Post-dose | 0.2 (6.32) | -0.8 (5.88) | 7.2 (8.94) | 0.1 (4.51)
  16 Hour Post-dose | 3.6 (8.14) | 3.8 (7.79) | 9.6 (6.99) | 3.7 (6.89)
  24 Hour Post-dose | -3.8 (8.18) | -4.1 (6.16) | 0.9 (6.97) | -4.9 (6.05)

21. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: QTcP Interval
Description: The effect of evobrutinib on baseline-corrected measurements of QTcP was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: as for outcome 17
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
milliseconds
  Baseline | 388.2 (17.69) | 387.5 (17.40) | 389.1 (17.18) | 388.9 (17.08)
  15 Minutes Post-dose | 1.9 (5.21) | 2.1 (5.54) | -0.1 (4.06) | 3.2 (3.71)
  30 Minutes Post-dose | 0.8 (5.51) | 0.1 (4.57) | 2.5 (6.65) | 1.9 (4.32)
  1 Hour Post-dose | -0.6 (4.91) | -0.3 (5.15) | 9.8 (7.30) | 2.5 (5.47)
  1.5 Hour Post-dose | -3.1 (4.95) | -3.4 (5.18) | 10.9 (8.35) | 1.7 (5.45)
  2 Hour Post-dose | -2.4 (4.06) | -3.1 (3.94) | 13.0 (8.26) | -0.1 (5.33)
  2.5 Hour Post-dose | -3.1 (5.59) | -3.7 (5.20) | 10.7 (6.57) | -1.3 (4.45)
  3 Hour Post-dose | -3.7 (6.33) | -3.5 (4.60) | 11.7 (5.43) | -1.2 (5.18)
  4 Hour Post-dose | -2.9 (5.43) | -2.0 (5.71) | 9.4 (6.86) | -1.0 (5.65)
  6 Hour Post-dose | -2.6 (7.96) | -1.7 (7.46) | 5.8 (8.54) | -0.0 (7.63)
  8 Hour Post-dose | -3.0 (6.12) | -5.2 (7.82) | 6.3 (8.36) | -1.4 (8.29)
  12 Hour Post-dose | 0.8 (6.20) | -0.9 (5.90) | 8.2 (9.62) | 0.3 (4.98)
  16 Hour Post-dose | 4.9 (8.65) | 4.5 (8.10) | 11.3 (7.53) | 5.8 (7.07)
  24 Hour Post-dose | -1.5 (8.22) | -3.2 (6.86) | 2.5 (7.33) | -2.9 (6.47)

22. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: PR Interval
Description: The effect of evobrutinib on baseline-corrected measurements of PR interval was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: as for outcome 17
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
milliseconds
  Baseline | 166.7 (16.59) | 170.4 (17.93) | 167.7 (17.73) | 167.1 (17.99)
  15 Minutes Post-dose | -0.2 (4.66) | -1.2 (5.29) | -0.8 (4.01) | -1.3 (4.36)
  30 Minutes Post-dose | 0.5 (3.72) | 2.6 (4.37) | -1.2 (5.27) | 0.1 (5.14)
  1 Hour Post-dose | 1.1 (4.13) | 1.2 (4.04) | -1.5 (7.52) | -0.8 (5.11)
  1.5 Hour Post-dose | 1.9 (5.11) | 0.9 (5.15) | -1.9 (7.41) | -0.9 (5.69)
  2 Hour Post-dose | 0.9 (4.91) | -0.5 (3.59) | -2.5 (8.15) | -0.3 (5.24)
  2.5 Hour Post-dose | 0.6 (4.64) | -1.8 (5.20) | -3.5 (6.49) | -1.4 (6.69)
  3 Hour Post-dose | 0.1 (5.69) | -1.5 (5.45) | -3.7 (7.42) | -3.0 (5.16)
  4 Hour Post-dose | -0.5 (7.11) | -1.2 (5.01) | -3.6 (7.77) | -4.2 (4.16)
  6 Hour Post-dose | -9.3 (7.52) | -9.4 (4.73) | -10.6 (8.22) | -11.1 (8.48)
  8 Hour Post-dose | -8.3 (6.98) | -9.3 (6.53) | -9.3 (7.30) | -11.1 (7.17)
  12 Hour Post-dose | -2.2 (7.43) | -3.9 (8.28) | -3.6 (8.03) | -2.8 (6.28)
  16 Hour Post-dose | -2.6 (8.70) | -5.2 (7.20) | -3.1 (7.95) | -4.1 (6.25)
  24 Hour Post-dose | -1.0 (7.00) | -2.6 (6.14) | -0.5 (9.38) | -1.2 (7.99)

23. Secondary Outcome: Effect of Evobrutinib on ECG Parameters: QRS Duration
Description: The effect of evobrutinib on baseline-corrected measurements of QRS duration was summarized by treatment and time points using descriptive statistics. Absolute change from baseline values was reported.
Time Frame: as for outcome 17
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Evobrutinib 45mg | Evobrutinib 225mg | Moxifloxacin 400mg | Placebo
Number analyzed (Participants) | 31 | 32 | 32 | 32
milliseconds
  Baseline | 91.7 (8.28) | 91.8 (8.24) | 91.7 (8.11) | 91.0 (8.12)
  15 Minutes Post-dose | 0.1 (1.44) | 0.3 (1.15) | 0.1 (1.31) | 0.4 (1.23)
  30 Minutes Post-dose | 0.4 (1.25) | 0.4 (1.41) | -0.4 (1.22) | 0.7 (1.44)
  1 Hour Post-dose | -0.1 (1.20) | 0.4 (1.02) | 0.2 (1.26) | 0.5 (1.29)
  1.5 Hour Post-dose | -0.4 (1.30) | -0.2 (1.29) | -0.1 (1.16) | -0.1 (1.15)
  2 Hour Post-dose | -0.5 (1.17) | -0.6 (1.47) | -0.1 (1.42) | -0.5 (1.60)
  2.5 Hour Post-dose | -0.6 (1.29) | -0.3 (1.64) | -0.2 (1.27) | -0.3 (1.59)
  3 Hour Post-dose | -0.5 (1.35) | -0.1 (1.50) | -0.1 (1.03) | -0.1 (1.35)
  4 Hour Post-dose | -0.7 (1.41) | -0.3 (1.71) | -0.4 (1.70) | 0.0 (1.53)
  6 Hour Post-dose | -0.6 (2.26) | -0.5 (2.12) | -0.6 (1.70) | -0.4 (1.98)
  8 Hour Post-dose | -0.8 (1.99) | -0.5 (1.78) | -0.1 (1.82) | 0.4 (1.97)
  12 Hour Post-dose | -0.2 (1.95) | 0.2 (2.14) | 0.2 (1.45) | 0.2 (1.85)
  16 Hour Post-dose | 0.0 (1.91) | 0.4 (1.74) | 0.6 (1.90) | 0.8 (2.08)
  24 Hour Post-dose | 0.5 (1.93) | 0.1 (1.22) | 0.3 (1.31) | 0.5 (1.43)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Groups:
- 400 mg Moxifloxacin: Participants received single oral dose of Moxifloxacin 400mg in treatment period 1, 2, 3 or 4under fasted condition
- 45 mg Evobrutinib: Participants received single oral dose of Evobrutinib 45 milligram (mg) in treatment period 1, 2, 3 or 4 under fasted condition
- 225 mg Evobrutinib: Participants received single oral dose of Evobrutinib 225 mg in treatment period 1, 2, 3 or 4 under fasted condition
Arm/Group | Placebo | 400 mg Moxifloxacin | 45 mg Evobrutinib | 225 mg Evobrutinib
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 8/32 | 5/32 | 8/31 | 5/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | 400 mg Moxifloxacin (N=32) | 45 mg Evobrutinib (N=31) | 225 mg Evobrutinib (N=32)
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT07214935/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT07214935/SAP_001.pdf